CLINICAL TRIAL: NCT04039789
Title: Impact of Physical Activity as a Coadjuvant Treatment in the Healing of Venous Ulcers in Primary Health Care: Multicenter Randomized Clinical Trial - Active Legs Project
Brief Title: Impact of Physical Activity as a Coadjuvant Treatment in the Healing of Venous Ulcers in Primary Health Care.
Acronym: ACTIVE_LEGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Principal Investigator, Borja Jesús Herraiz Ahijado, Principal Investigator. Clinical nurse, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCI 11/18
Record Dates: First submitted 2019-07-11; First posted 2019-07-31 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Varicose Ulcer
Keywords: Varicose ulcer; Exercise; Nurses; Healthy Aging
MeSH Terms: conditions — Varicose Ulcer; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised, multicentre clinical trial, parallel, pragmatic, with 6 months of follow-up.
Masking Description: Intervention can't be masked. We will objectify primary outcome by photography images and adherence to exercise through the use of pedometers.
  Statistician conducting the analysis will not know to which study arm a given patient has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Usual Care: that consists of healing the wound (assessment, cleaning, disinfection, debridement and topical treatment) and compression therapy multilayer usual practice, according to the recommendations for the treatment of cutaneous ulcers of the Region of Madrid.
  Interventions: Procedure: Usual care
- Intervention (Experimental): ACTIVE LEGS: The usual care plus experimental intervention. It is a structured educational intervention, directed by nurses and carried out in the health center consultations. The intervention "Active Legs" has been designed based on the available evidence. It incorporates a program of lower limb exercise at home and daily walking patterns.
  Home program of lower limb exercises. The nurse will instruct the patients in the performance of 4 exercises of lower limbs of progressive difficulty that must be performed at home 5 days a week, twice a day Daily walking program. In addition, patients must ambulate progressively until reaching the marked goal (150 min / week (30 minutes for 5 days a week)) .
  At the start of the study, the "Active Legs" diary will be provided, showing the patterns of the exercise and walking program graphically and a pedometer.
  Interventions: Behavioral: Project active legs; Procedure: Usual care

INTERVENTIONS:
Behavioral: Project active legs — Home program of exercises of lower extremities includes the performance of 4 exercises of lower extremities of progressive difficulty that must be carried out at home 5 days a week, twice a day and walking progressively until reaching the marked goal (150 min / week (30 minutes for 5 days a week)).
  Arms: Intervention
Procedure: Usual care — Evaluation, cleaning, debridement, topical treatment (moist healing) and compressive therapy according to the recommendations for the treatment of chronic cutaneous ulcers of the Community of Madrid.

SUMMARY:
Objectives: To evaluate the effectiveness of a structured educational intervention in physical exercise "Active Legs" as an adjuvant treatment to improve the healing of chronic venous ulcers at 3 months of follow-up, compared with the usual practice in people treated in primary care. Secondary objectives: To evaluate if the intervention active legs as an adjuvant treatment produces better results than usual practice in: degree of healing, recurrence, complete healing at 6 months, pain and quality of life. Describe degree of adherence and satisfaction with the intervention. Design: Randomized, multicenter, pragmatic, open clinical trial of parallel groups with 6 months of follow-up. Setting: Primary Care Health Centers (Madrid). Subjects: Patients with venous ulcers, with treatment in the nursing consultation of the participating centers. Sample: 224 participants (112 in each group). Intervention: Both groups will receive the usual treatment of cleaning, debridement based on humid environment cure and multilayer compression therapy according to the recommendations of Community of Madrid. The intervention group will also receive the structured educational intervention of lower limbs physical exercise and daily walking patterns. Variables: Main: complete healing at 3 months follow-up. Secondary: Degree of healing; ulcer area; quality of life; pain, related to the healing process, prognosis and recurrences; Sociodemographic and related adherence and satisfaction. Data analysis: Main effectiveness: comparison of the incidence of ulcers with complete healing at 3 months of follow-up in both groups, time to complete healing (Kaplan-Meier and Log-rank test). Adjustment of prognostic factors (Cox regression).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of venous ulcers registered in electronic clinical history (history of chronic venous insufficiency and/or venous ulcer) and presence of an ankle brachial index (ABI) greater than 0.8 and less than 1.3.
* Presence at least a venous ulcer of 1cm or more in diameter. If the participant has more than one lesion, the nurse will select the lesion with the highest Resvech 2.0 score for the study.
* Independent ambulation or with the help of devices.
* Individuals who able to follow the demands of the trial and who provide their written informed consent to participate.

Exclusion Criteria:

* Patients with mixed ulcers.
* Acute phase deep vein thrombosis.
* Patients on treatment with antineoplastic agents.
* Decompensated heart failure.
* Rheumatoid arthritis.
* Acute phase dermatitis, at the time of the study.
* Patients immobilized at home, institutionalized or displaced residing outside the area where the research is conducted for more than 6 months a year or during the performance of the intervention.
* Absolute contraindication to perform physical exercise.
* Patients who are simultaneously participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Complete healing at 6 months of follow-up | 6 months
  (yes/no) (complete and sustained epithelialisation for at least 2 weeks).
Time elapsed between start of the study and complete healing of the wound | 6 months
  (in days)

SECONDARY OUTCOMES:
Degree of healing (Resvech 2.0) | Measured at the beginning (basal) and fortnightly up to 3 months and at 6 months.
  The questionnaire consists of 6 dimensions with ascending scoring scales according to the severity of the dimension studied. It is divided into: depth (0 to 4), size (0 to 6), borders (0 to 4), wound bed (0 to 4), exudate (0 to 3) and signs and symptoms of infection (0 to 14). The total score ranges from 0 to 35.
Ulceral area | Measured at the beginning (basal) and fortnightly up to 3 months and at 6 months.
  In cm2. Measured by digital photography. Measurement through digital photography and subsequent treatment of the image using the open source Java image processing program "The ImageJ ecosystem" and its subsequent calculation using the Visitrack device.
Health-related quality of life for patients with venous ulcers (CCVUQ-e) | Measured at the beginning (baseline), in the middle (3 months) and at the end of the study (6 months).
  It is a questionnaire that measures quality of life in patients with venous ulcers. In addition to a global synthetic quality of life score, it has 4 dimensions: Social interaction, Cosmesis (body image), Emotional state and Domestic activities. Both the general score and the dimensions have a score that ranges from 0 to 100, where 0 is the best quality of life and 100 the worst quality of life.
Perceived pain: visual analogical scale of the McGill questionnaire | Measured at the beginning (baseline), in the middle (3 months) and at the end of the study (6 months).
  The visual analogical scale of the McGill questionnaire will be used. A greater than 20mm in the Visual Analog Scale of pain scale will be considered a clinically significant change.
  It goes from "no pain" 0 to "unbearable pain" 10, the patient will mark that point on the line that best reflects the pain he suffers.
Level of adherence to the intervention "Active Legs". Number of steps. | In the intervention group. Measured biweekly coinciding with follow-up visits up to 3 months and 6 months.
  Daily record using the Yamax PZ270 pedometer (15 days memory)
Level of adherence to the intervention "Active Legs". Time. | In the intervention group. Measured biweekly coinciding with follow-up visits up to 3 months and 6 months.
  The time in minutes / day
Level of adherence to the intervention "Active Legs". The self-reported information by the patient of the domiciliary exercise program. | In the intervention group. Measured biweekly coinciding with follow-up visits up to 3 months and 6 months.
  By registering in the activity diary, classifying it as "Excellent" in 75% or more of the prescribed sessions, "Good" between 50-74%, "Moderate" between 25-49% and "Poor" less than 25%.
Age (sociodemographic variables) | Measured at the beginning (baseline)
  in years
Sex (sociodemographic variables) | Measured at the beginning (baseline)
  Male/Female
Living alone (sociodemographic variables) | Measured at the beginning (baseline)
  Yes/no
Employment status (sociodemographic variables) | Measured at the beginning (baseline)
  housewife / unemployed / student / worker employee account / worker own account
Education level (sociodemographic variables) | Measured at the beginning (baseline)
  low / medium / high
Weight (variables related to the healing process) | Measured at the beginning (baseline)
  in kilograms. weight and height will be combined to report BMI in kg/m^2
Height (variables related to the healing process) | Measured at the beginning (baseline)
  in meters. weight and height will be combined to report BMI in kg/m^2
Underlying disease (variables related to the healing process) | Measured at the beginning (baseline)
  (yes / no) for heart failure, renal failure, hypertension, diabetes mellitus, rheumatoid arthritis, asthma, chronic obstructive pulmonary disease, osteoarthritis, deep vein thrombosis, peripheral arterial vasculopathy, varicose veins.
ABI (variables related to the healing process) | Measured at the beginning (baseline)
  The Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm. It has been shown to be a specific and sensitive metric for the diagnosis of Peripheral Arterial Disease (PAD).
Tobacco consumption (variables related to the healing process) | Measured at the beginning (baseline)
  no smoker / smoker / ex-smoker
Alcohol consumption (variables related to the healing process) | Measured at the beginning (baseline)
  volume grams of alcohol / week
Topical and systemic treatment (variables related to the healing process) | Measured at the beginning (baseline)
  (yes/no) for hydrocellular dressings, alginates, hydrogels, collagenase, silver dressings, low adhesion dressings, silver sulfadiazine in ointment, other antibiotics in ointment, moisturizing products for the skin.
Adherence to multilayer compression therapy (variables related to the healing process) | Measured at the beginning (basal) and fortnightly until 3 months and at 6 months .
  (yes/no)
Physical activity level measured by the Minnesota free time physical activity questionnaire (variables related to the healing process) | Measured at the beginning (baseline), in the middle (3 months) and at the end of the study (6 months).
  It allows to measure the energy expenditure during free time and allows to classify individuals in activity categories. In metabolic energy turnover (METS)-min/14 days. Interpreting as: very active above 5000 METS-min / 14 days, Active between 3000 and 4999 METS-min / 14 days, Moderately active between 1250 and 2999 METS-min / 14 days and sedentary less than 1250 METS-min / 14 days .
Type of daily walking (variables related to the healing process) | Measured at the beginning (baseline)
  Independent / Independent with technical assistance (cane, crutches or walker with or without wheels) / With the help of the participation of a person without technical assistance / With the help of the participation of a person with technical help
Location of the ulcer (prognostic variables) | Measured at the beginning (baseline)
  internal lateral aspect/ supra-malleolar area/ anterior area of the leg/ external lateral aspect of the leg/ posterior aspect of the leg
Number of ulcers at the time of the study (prognostic variables) | Measured at the beginning (baseline)
  in number
Time in days of evolution of the venous ulcers before inclusion in the study (prognostic variables) | Measured at the beginning (baseline)
  in days
Recurrent ulcer (prognostic variables) | Measured at the beginning (baseline)
  (yes/no)
Recurrence (variables related to recurrences) | measured at 6 months of follow-up
  (yes / no)
Use of compression stockings (variables related to recurrences) | measured at 6 months of follow-up
  (Yes/no) for Light / normal / strong compression
Hydration of the legs (variables related to recurrences) | measured at 6 months of follow-up
  (Yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Borja Jesús Herraiz Ahijado, Nurse, Principal Investigator — Gerencia Asistencial de Atención Primaria de la Comunidad de Madrid
Locations (1):
- Borja Jesús Herraiz Ahijado, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herraiz-Ahijado B, Folguera-Alvarez C, Rodriguez-Barrientos R, Sanchez-Ruano R, Pascual-Garcia M, Mori-Vara P, Verdu-Soriano J, Rico-Blazquez M; Active Legs Group. Impact of physical activity as an adjuvant treatment in the healing of venous ulcers in primary care: active legs RCT. BMC Nurs. 2025 Dec 10;25(1):38. doi: 10.1186/s12912-025-04189-0. PMID 41372918
- [Derived] Herraiz-Ahijado B, Folguera-Alvarez C, Verdu-Soriano J, Mori-Vara P, Rico-Blazquez M. Active legs: Impact of physical activity as an adjuvant treatment in the healing of venous ulcers in primary care: a RCT protocol study. BMC Nurs. 2023 Mar 10;22(1):65. doi: 10.1186/s12912-023-01214-y. PMID 36899351